CLINICAL TRIAL: NCT05990816
Title: Natural Course of Homocysteine After Uneventful Total Joint Arthroplasty
Status: Not yet recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Cemil Burak DEMİRKIRAN, Resident Doctor, Bezmialem Vakif University
Other Study IDs: cbdemirkan
Record Dates: First submitted 2023-08-05; First posted 2023-08-14 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Joint Prosthesis; Complications, Infection or Inflammation
Keywords: periprosthetic joint infection; diagnosis; natural course; total joint arthroplasty.
MeSH Terms: conditions — Infections; Inflammation; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Test for Homocysteine Levels Assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arthroplasty Patients: Only one group that consist patients who underwent primary total joint arthroplasty
  Interventions: Diagnostic Test: Blood works for homocysteine levels

INTERVENTIONS:
Diagnostic Test: Blood works for homocysteine levels — In a single patient group of 80 people, the natural course of homocysteine after total joint arthroplasty will be examined by blood work analyzes at the 1,2,3,4 and 6th weeks after operation

SUMMARY:
The goal of this observational study is to asses the natural course of blood homocysteine levels in patients who underwent primary total joint arthroplasty surgery. The main question[s] it aims to answer are:

* İs homocysteine a good marker for determining periprosthetic joint infection ?
* İs homocysteine more sensitive marker for periprosthetic joint infections ?

ELIGIBILITY:
Inclusion Criteria:

* People who have undergone Total Knee Arthroplasty operation
* People who have undergone Total Hip Arthroplasty operation

Exclusion Criteria:

* People who have undergone total knee arthroplasty operation and developed a periprosthetic joint infection
* People who have undergone total hip arthroplasty operation and developed a periprosthetic joint infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healty volunteers who have undergone uneventful primary total joint arthroplasty
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Homocysteine | 6 months
  Homocysteine levels in patient blood works

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Mouravas H, Verettas D, Kazakos K, Xarhas K, Panagiotou N, Ellinas P. Homocysteine and its relationship to deep venous thrombosis in patients undergoing total knee or hip arthroplasty. Hippokratia. 2010 Jul;14(3):185-8. PMID 20981167
- [Background] Watanabe N, Ogawa T, Takada R, Amano Y, Jinno T, Koga H, Yoshii T, Okawa A, Miyatake K. Association of osteoporosis and high serum homocysteine levels with intraoperative periprosthetic fracture during total hip arthroplasty: a propensity-score matching analysis. Arch Orthop Trauma Surg. 2023 Dec;143(12):7219-7227. doi: 10.1007/s00402-023-04989-6. Epub 2023 Jul 19. PMID 37468711
- [Result] Azboy I, Catal B, Basarir K, Mutlu M, Bilgen OF, Parvizi J. The Natural Course of Serum D-Dimer, C-Reactive Protein, and Erythrocyte Sedimentation Rate Levels After Uneventful Primary Total Joint Arthroplasty. J Arthroplasty. 2021 Sep;36(9):3118-3122. doi: 10.1016/j.arth.2021.04.031. Epub 2021 Apr 30. PMID 34088567